CLINICAL TRIAL: NCT00600665
Title: Computerized PAINRelieveIt for Adult Sickle Cell Disease
Brief Title: Effectiveness of a Computerized Tool (PAINRelieveIt) to Help Manage Pain Related to Sickle Cell Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Diana J. Wilkie, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 420; R01HL078536 (NIH)
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Anemia, Sickle Cell; Hemoglobin SC Disease
Keywords: Sickle Cell Anemia; Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell; Hemoglobin SC Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (Active Comparator): In Part 1 of the study, participants will access PAINReportIt and computer games. PAINReportIt helps the patient describe the pain experienced. In Part 2 of the study, participants will continue to access PAINReportIt when they are seen in the clinic, emergency department (ED), acute care center (ACCA), and hospital. They will gain access to the PAINUCope computer-based programs, which provides multimedia education tailored to the patient's misconceptions about pain management. They will receive medial usual care at the outpatient clinic, ED, ACC, and hospital.
  Interventions: Behavioral: PAINReportIt; Behavioral: PAINUCope
- PAINUCope/PAINConsultN (Experimental): In Part 1 of the study, participants will access PAINReportIt and PAINUCope computer-based programs. PAINReportIt helps the patients describe the pain experiences and PAINUCope provides multimedia education tailored to the patient's misconceptions about pain management. In Part 2 of the study, participants will continue to access PAINReportIt and PAINUCope programs when they are seen in the clinic, emergency department (ED), acute care center (ACC), and hospital. Their doctors will have access to PAINConsultN when seen at the ED, ACC, and hospital. PAINConsultN is just-in-time decision support for the physicians with the pain data summarized and suggestions for analgesics that may be useful to help manage the patient's pain.
  Interventions: Behavioral: PAINReportIt; Behavioral: PAINUCope; Behavioral: PAINConsultN

INTERVENTIONS:
Behavioral: PAINReportIt — A pain assessment data collection tool
Behavioral: PAINUCope — A multimedia patient education program tailored to the participant's SCD pain management misconceptions
Behavioral: PAINConsultN — A decision support tool for doctors that will provide algorithm-based pain medication therapies tailored to each participant's pain level
  Arms: PAINUCope/PAINConsultN

SUMMARY:
Sickle cell disease (SCD) is a blood disorder that is characterized by intense, painful episodes known as sickle cell crises. This study will evaluate the effectiveness of PAINRelieveIt, a three-part computer-based pain management tool, in treating adults with SCD.

DETAILED DESCRIPTION:
SCD is an inherited blood disorder that mainly affects people of African, Mediterranean, or Latin descent. Symptoms include anemia, infections, organ damage, and painful sickle cell crises. Adults with SCD who experience frequent painful crises are more likely to die sooner than are adults with SCD who have fewer painful crises. Experts suggest that SCD pain be treated in the same way that cancer pain is treated because both types of pain are sustained and severe. However, unlike the research directed towards cancer pain, research focused on the characteristics of SCD pain has been limited. Although medications are available to treat SCD pain, the SCD pain management process is complex and often requires more time than what is available during the typical medical appointment. Recent advances in computer technologies may provide an opportunity to improve the effectiveness of SCD pain management by combining online patient education with decision-making support tools for doctors. This study will evaluate three touch screen computerized tools that are known collectively as PAINRelieveIt. The three tools include the following:

1. PAINReportIt-a pain assessment data collection tool
2. PAINUCope-a multimedia patient education program tailored to the participant's SCD pain management misconceptions
3. PAINConsultN-a decision support tool for doctors that will provide algorithm-based pain medication therapies tailored to each participant's pain level

This two-part study will evaluate the effectiveness of PAINReportIt and PAINUCope, alone and in combination with PAINConsultN, at improving participants' SCD pain by educating participants about their role in pain management and by providing decision-making support to doctors.

This study comprises two parts. Part 1 of the study will enroll patients who are receiving care at the University of Illinois at Chicago Sickle Cell Clinic. The patients will be randomly assigned to receive 3 months of either access to PAINReportIt and PAINUCope or usual care. At baseline and Month 3, participants will complete questionnaires on misconceptions about pain, medication adherence, and pain intensity. The same participants from Part 1 of the study will be enrolled into Part 2 of the study, which will last 2 years. Part 2 participants will be randomly assigned to receive either care from doctors who have access to PAINConsultN or usual care. All participants will have access to PAINReportIt and PAINUCope. At baseline and Year 2, participants will complete questionnaires on pain episodes. Information will also be collected from doctors, including pain documentation, appropriateness of prescribed pain medications, and the number of emergency department visits by and hospitalizations of participants experiencing painful SCD crises.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with SCD
* Scheduled for continuing care at the University of Illinois at Chicago Sickle Cell Clinic
* Experienced a moderate to severe level of pain (at least 3 on 0 to 10 scale) related to the SCD within the 12 months prior to study entry
* Had a emergency department visit or hospitalization within the 2 years prior to study entry
* Speaks and reads English

Exclusion Criteria:

* Legally blind
* Physically unable to complete study questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2007-02; Primary Completion 2013-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
For Part 1 of the study: misconceptions about pain, analgesic adherence, and pain intensity measured by the composite pain index (CPI) | Measured at Month 3
For Part 2 of the study: number of participant-reported pain episodes, pain documentation and appropriateness of prescribed analgesics as measured by doctors, and number of emergency department visits and hospitalizations | Measured at Year 2

CONTACTS AND LOCATIONS:
Overall Officials: Diana J. Wilkie, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago Sickle Cell Center and Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Result] Wilkie DJ, Molokie R, Boyd-Seal D, Suarez ML, Kim YO, Zong S, Wittert H, Zhao Z, Saunthararajah Y, Wang ZJ. Patient-reported outcomes: descriptors of nociceptive and neuropathic pain and barriers to effective pain management in adult outpatients with sickle cell disease. J Natl Med Assoc. 2010 Jan;102(1):18-27. doi: 10.1016/s0027-9684(15)30471-5. PMID 20158132